CLINICAL TRIAL: NCT04880525
Title: The Effect of a Weight-Loss Diet in Women Doing Reformer Pilates: A 12-Week Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Çağla AYER, Research Assistant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-629
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Pilates; Diet; Women
Keywords: Pilates-based exercises; Weight Loss; Diet; Women; Body composition
MeSH Terms: conditions — Weight Loss | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: For a period of 12 weeks, subjects in the Study Group (SG) and Control Group (CG) groups received three 45-minute sessions of Pilates exercises per week.
  Study Group: In addition to Pilates, she followed a three-month weight-loss diet based on Turkey Dietary Guidelines, as prescribed by the dietician. These diet plans were designed to ensure that carbohydrates provided 45-60% of the energy, protein provided 10-20%, and fat provided 20-35 percent.
  Control Group: The women in the control group did only reformer pilates for three months. They were followed up for not applying any diet.
Masking Description: There was no masking in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The study group does reformer pilates for 45 minutes 3 days a week. The intensity of the workouts was gradually increased. Warm-up (10 minutes), main Pilates training activity (25 minutes), and cool-down (10 minutes) were the three parts of each session (10 minutes). In addition to pilates, the women in the SG followed a personalized weight loss diet. In accordance with Turkey Dietary Guidelines, these diet plans were designed to provide 45-60% of energy from carbohydrates, 10-20% from protein, and 20-35 percent from fat.
  Interventions: Other: Dietary intervention
- Control Group (No Intervention): The control group does reformer pilates for 45 minutes 3 days a week. The intensity of the workouts was gradually increased. Warm-up (10 minutes), main Pilates training activity (25 minutes), and cool-down (10 minutes) were the three parts of each session (10 minutes). Individuals in the CG received no dietary or nutritional intervention. On any diet, the status of women in the CG was frequently questioned.

INTERVENTIONS:
Other: Dietary intervention — In accordance with Turkey Dietary Guidelines, these diet plans were designed to provide 45-60% of energy from carbohydrates, 10-20% from protein, and 20-35 percent from fat.
  Arms: Study Group

SUMMARY:
The purpose of this study is to determine the effect of a weight-loss diet on body composition in women who practice reformer pilates for 12 weeks. It compares dietary habits and macro and micronutrient intakes in subjects with and without a weight-loss diet at the start and end of the study.

DETAILED DESCRIPTION:
The effect of a weight-loss diet on body composition in women reformer pilates for 12 weeks was compared in this study. It compares dietary habits and macro and micronutrient intakes in subjects with and without a weight-loss diet at the start and end of the study.

A total of 49 women (18 years old) were randomly assigned to one of two groups: control (CG: reformer pilates; n=23) or study (SG: reformer pilates + weight-loss diet; n=26). Subjects in both groups did pilates for 45 minutes three times a week for a total of 12 weeks. At the start and end of the study, their body weight (kg), waist circumference (cm), hip circumference (cm), neck circumference (cm), mid-upper arm circumference (cm), and body composition [body fat (% ), body water (% ), body muscle (% )] were all measured. Their waist/height ratio and body mass index (kg/m2) were also measured at the start and end of the study. All subjects' dietary habits were questioned, their 24-hour retrospective food consumption was recorded, and their physical activity levels were assessed using the International Physical Activity Questionnaire (Short Form).

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study
* Being in the age range of 18-65
* Female
* Not a regular Pilates practitioner, and physically independent to perform basic daily activities

Exclusion Criteria:

* Refuse to participate in the study
* Being younger than 18 or over 65
* Male
* A regular Pilates practitioner
* Not being suitable for physical activity

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — It became well-known in the twentieth century, particularly among women. Reformer pilates exercises are preferred by women for aesthetic reasons such as weight loss, slimming, staying in shape, muscle strengthening, muscle pain relief, and flexibility.
Enrollment: 49 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in anthropometric measurements | 12 weeks
  At the start and end of the study, their body weight (kg), waist circumference (cm), hip circumference (cm), neck circumference (cm) and mid-upper arm circumference (cm) were all measured. These measurements are expected to change according to the beginning of the study.
Change in body composition | 12 weeks
  At the start and end of the study, their body fat (%), body water (%), body muscle (%) were all measured. Their waist-to-height ratio and body mass index (kg/m2) were also measured at the beginning and end of the study. These measurements are expected to change according to the beginning of the study.
Food consumption | 12 weeks
  Their 24-hour retrospective food consumption were taken
Physical activity levels | 12 weeks
  Their physical activity levels were evaluated through the International Physical Activity Questionnaire (IPAQ Short Form). This form had seven questions and asked about the amount of time spent sitting, walking, moderate, and vigorous activities. The total score accounted for the duration (minutes) and frequency (days) of the activities completed. Physical inactivity (600 MET -min/week), low physical activity (600-3000 MET -min/week), and adequate physical activity (with health benefits) (>3000 MET -min/week) were defined.

CONTACTS AND LOCATIONS:
Overall Officials: Çağla Ayer, M.D., Principal Investigator — Izmir Katip Çelebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Cigli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study's data is planned to be published and shared in a scientific paper